CLINICAL TRIAL: NCT03441373
Title: Clinical Study to Assess Efficacy, Safety, Tolerability and Optimal Dose Ranging of XC8 in Doses 20, 100 and 200 mg Once Daily in Patients With Uncomplicated Influenza or Other Acute Respiratory Viral Infections (ARVI)
Brief Title: XC8 in the Treatment of Patients With Acute Respiratory Viral Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLU-XC8-01
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Influenza; Acute Respiratory Infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- XC8 20 mg and Placebo (Group A) (Experimental): XC8 20 mg orally. 2 tablets of XC8 10 mg +2 tablets of Placebo 100 mg (in total 4 tablets) once daily during 5 days of treatment period
  Interventions: Drug: XC8 20 mg
- XC8 100 mg and Placebo (Group B) (Experimental): XC8 100 mg orally.
  1 tablet of XC8 100 mg +2 tablets of Placebo 10 mg + 1 tablet of Placebo 100 mg (in total 4 tablets) once daily during 5 days of treatment period
  Interventions: Drug: XC8 100 mg
- XC8 200 mg and Placebo (Group C) (Experimental): XC8 200 mg orally. 2 tablets of XC8 100 mg +2 tablets of Placebo 10 mg (in total 4 tablets) once daily during 5 days of treatment period.
  Interventions: Drug: XC8 200 mg
- Placebo (Group D) (Placebo Comparator): Placebo orally.
  Interventions: Drug: XC8 20 mg; Drug: XC8 100 mg; Drug: XC8 200 mg; Drug: Placebo

INTERVENTIONS:
Drug: XC8 20 mg — once daily during 5 days.
  Other Names: Нistamine glutarimide
  Arms: Placebo (Group D); XC8 20 mg and Placebo (Group A)
Drug: XC8 100 mg — once daily during 5 days.
  Other Names: Нistamine glutarimide
  Arms: Placebo (Group D); XC8 100 mg and Placebo (Group B)
Drug: XC8 200 mg — once daily during 5 days.
  Other Names: Нistamine glutarimide
  Arms: Placebo (Group D); XC8 200 mg and Placebo (Group C)
Drug: Placebo — once daily during 5 days.
  Arms: Placebo (Group D)

SUMMARY:
A multicenter double-blind, randomized, placebo-controlled, parallel-group comparative Phase II / III clinical study to assess safety, tolerability, efficacy and optimal dose ranging of XC8 vs. placebo in patients with uncomplicated influenza or other ARVI during a 5-day treatment.

The primary objective of the study was to demonstrate the difference in time before the onset of a sustained improvement in clinical symptoms according to the Severity Rating Scale for ARVI, and to determine the optimal dose of XC8 in the treatment of influenza and other ARVI.

DETAILED DESCRIPTION:
Twenty-three Russian centers were approved for participation in this study. Twenty centers were initiated. Patients were enrolled in 18 centers. The study consisted of two parts: phase II and phase III. Each of the parts included 3 periods: screening, treatment, follow-up.

In the first part of the study (Phase II), all eligible patients were randomized into 4 groups (groups A, B, C, and D) in a 1:1:1:1 ratio:

Group A - XC8 20 mg daily (40 patients); Group B - XC8 100 mg daily (40 patients); Group C - XC8 200 mg daily (40 patients); Group D - placebo (40 patients).

Interim analysis was planned after the end of the first part of the study (Phase II). Based on the results of the interim analysis, the most promising XC8 dose group was selected and the necessary set was calculated to compare this group with the placebo group by the primary endpoint in a pooled set using an adaptive design with type I error control.

In the second part of the study (Phase III), all eligible patients were randomized into 2 groups (groups C and D) in a 1:1 ratio:

Group C - XC8 200 mg daily (80 patients); Group D - placebo (80 Patients).

During the treatment period (5 days), patients received XC8 / placebo daily on a background of standard symptomatic therapy. The follow-up period lasted for 9 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 45 years (inclusively).
2. Clinically diagnosed influenza or other acute or moderate ARVI based on the patient's body temperature ≥37.5ºС, nasal congestion or profuse rhinorrhea and at least 1 of the following symptoms of intoxication: headache, general malaise, myalgia, pain in the eyeballs.
3. Uncomplicated course of ARVI or influenza.
4. The onset of symptoms no more than 36h prior to the inclusion into the study.
5. Women of reproductive age (who are not in menopause and who have not undergone surgical sterilization) and men who have sexual activity should use a reliable method of contraception (acceptable methods of contraception in this study are: intrauterine devices, oral contraceptives, contraceptive patch, long-acting injectable contraceptives, a double barrier method (condom and diaphragm with spermicide) throughout the study period.
6. Compliance with the treatment regimen, visits and laboratory examinations provided by the protocol.
7. Signed Informant Consent Form.

Exclusion Criteria:

The patient will be deemed ineligible for the study meeting any of the following criteria:

1. Complicated course of influenza or ARVI (including the presence / development of bacterial infection).
2. Antiviral medications in 7 days prior to screening (antiviral agents, interferons and interferon inducers, drugs that have immunomodulating action) or anti-infective agents of systemic or local action.
3. Severe infection with signs of cardiovascular insufficiency development and other manifestations of infectious-toxic shock, as well as with the presence of neuroinfection syndrome (encephalic and meningoencephalic reactions, polyradiculoneuritis, neuritis).
4. Signs of the development of viral pneumonia (the presence of two or more of the following symptoms): dyspnea, chest pain when coughing, systemic cyanosis, dullness of percussion sound with a symmetrical evaluation of the upper and lower sections of the lungs).
5. Infectious diseases during the last week before including into the study.
6. History of bronchial asthma.
7. History of increased convulsive activity.
8. Severe, decompensated or unstable somatic diseases (any diseases or conditions that are life-threatening or may worsen the patient's prognosis, and make him/her ineligible for the clinical study).
9. History of oncological diseases, HIV, tuberculosis.
10. Hypersensitivity to excipients of the XC8.
11. Diabetes mellitus, lactose intolerance, lactase deficiency.
12. Drug or alcohol abuse.
13. Participation in any other clinical trial in the last 90 days.
14. Pregnancy or lactation.
15. Military or prison populations.
16. Impossibility or inability to comply with the study procedures.
17. A member of the investigator's family or other person interested in the results of the study
18. Abnormal laboratory results, which, according to the study doctor, interfere with the patient's inclusion in the study.
19. History of renal insufficiency.
20. Only for patients participating in Phase III study: Patient involvement in the first part of the study (Phase II) of FLU-XC8-01.

    -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Time to sustained improvement in clinical symptoms | up to Day 5
  Severity Rating Scale for ARVI (<2 points, provided that there is ≤ 1 point for one symptom) with temperature normalization (<37°C) (estimated by Kaplan-Meier), established according to patient diaries.

SECONDARY OUTCOMES:
Body temperature below 37°C without further elevation | up to Day 8
  Time to normalization of body temperature since the symptoms onset, measured in hours

CONTACTS AND LOCATIONS:
Locations (18):
- Russia (18):
  - Udmurt Republic Budgetary Healthcare Institution "City clinical Hospital #9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - State Educational Institution for further vocational education "Kazan State Medical Academy of Federal Healthcare Agency", Clinical site - State Independent Healthcare Institution "Republic Infectious Clinical Hospital n.a. professor Agafonov",, Kazan'
  - State Budgetary Institution of Higher Professional Education "Kuban State Medical University" of the Ministry of Health of the Russian Federation, Krasnodar
  - Nizhegorodsky region SBHI Nizhniy Novgorod Infectious Regional Clinical Hospital № 2, Nizhny Novgorod
  - Novosibirsk Municipal Healthcare Budgetary Institution "City Clinical Hospital # 19",, Novosibirsk
  - Novosibirsk region SBHI "City Infectious Clinical Hospital # 1",, Novosibirsk
  - ; Moscow region State Budgetary Institution "Podolsk City Clinical Hospital № 3", Podolsk
  - Municipal State Budgetary Institution "Rostov-on-Don City Clinical Hospital# 1 n.a. Semashko",, Rostov-on-Don
  - State Budgetary Institution of Higher Professional Education "Ryazan State Medical University n.a. Pavlov" of the Ministry of Health of the Russian Federation, Clinical site - SBHI of Ryazan region "Clinical Hospital n.a. Semashko", Ryazan
  - ArsVite Severo-Zapad LLC, Saint Petersburg
  - Federal State Budgetary institution "Diagnostic center with polyclinics" of the Administrative Department of the President of the Russian Federation, Saint Petersburg
  - Federal State Budgetary Institution "Research institute of influenza" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Saint Petersburg SHBI "City Clinical Hospital #40 of health resort administrative region", Saint Petersburg
  - Federal State Budgetary Institution Mordovia State Medical University n..a. N.P.Ogarev, Mordovia Republic SHBI "Republic Infectious Clinical Hospital", Saransk
  - State Budgetary Institution of Higher Professional Education "Siberian State Medical University" of the Ministry of Health of the Russian Federation, Tomsk
  - State Budgetary Institution of Higher Professional Education "Volgograd State Medical University" of the Ministry of Health of the Russian Federation, Clinical site - Infectious Regional Clinical Hospital № 1, Volgograd
  - State Budgetary Institution of Higher Professional Education "Yaroslavl State Medical University" of the Ministry of Health of the Russian Federation, Clinical site - Yaroslavl region State Healthcare Institution Infectious Regional Clinical Hospital # 1, Yaroslavl
  - State Budgetary Healthcare Institution (SBHI) of Yaroslavl region, Yaroslavl

IPD SHARING:
Plan to Share IPD: No